CLINICAL TRIAL: NCT02421562
Title: Training Nurses in Basic Hypnoanalgesia Techniques to Reduce Procedural Distress and Pain in Children: a Pilot Study
Brief Title: Training Nurses in Basic Hypnoanalgesia Techniques
Acronym: HYPNO-DIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Michel Duval, Dr Michel Duval, MD, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HYPNO-DIS
Record Dates: First submitted 2015-04-12; First posted 2015-04-20 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- training in hypnoanalgesia (Experimental): training nurses in hypnoanalgesia to perform painful procedure in children
  Interventions: Procedure: training in hypnoanalgesia

INTERVENTIONS:
Procedure: training in hypnoanalgesia — training nurses in hypnoanalgesia techniques to perform painful procedures in children followed in the outpatient hematology oncology clinic

SUMMARY:
Demonstrate that a 4-day training session will allow nurses to master basic hypnoanalgesia techniques, and this new tool will translate into a reduction of procedural distress and pain in their patients, thereby opening the way to larger clinical trials in various pediatric settings.

ELIGIBILITY:
Inclusion Criteria:

* children followed in the hematology-oncology outpatient clinic at least 4 times per year
* good understanding in French
* use of topic anesthesia or distraction object allowed, as long as used at all venipuncture measured sessions

Exclusion Criteria:

* prior use of hypnoanalgesia
* patients coming for emergency or non-scheduled appointment
* patients with acute pain on their scheduled appointment to the clinic
* acute psychiatric disease

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Practice performance of pediatric nurses after a 4-day training in hypnonalgesia techniques. Practice performance will be evaluated by two external evaluators on videotapes using a standardized scale. | 12 months

SECONDARY OUTCOMES:
Main secondary outcome measure : self-reported distress (fear) on VAS (visual analog scale). | 12 months
Distress evaluated with the Faces, Legs, Activity, Cry, Consolability scale by two external evaluators on video recordings. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michel Duval, MD, Principal Investigator — Ste-Justine Hospital
Locations (1):
- Ste-Justine Hospital, Montreal, Quebec, Canada